CLINICAL TRIAL: NCT03902821
Title: Reducing Overdose After Release From Incarceration
Acronym: ROAR
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Department of Corrections (Unknown); CODA Inc. (Unknown); Bridgeway Recovery (Unknown); Health Insight (Unknown); Oregon State University (Other)
Responsible Party: Principal Investigator, Elizabeth Waddell, Assistant Professor and Program Director, Oregon Health and Science University
Other Study IDs: ROAR
Record Dates: First submitted 2019-03-21; First posted 2019-04-04 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Overdose, Drug
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: XR-NTX and Certified Recovery Mentor — All consented participants will be offered an injection of extended-release naltrexone 3-7 days prior to release from prison. All consented participants will also be introduced to Certified Recovery Mentors one month prior to release.

SUMMARY:
The primary objective of the ROAR project is to evaluate an Oregon Department of Corrections (ODOC) pilot program that combines the use of extended-release naltrexone (XR-NTX) and Certified Recovery Mentors pre-release with linkage to community substance use disorder treatment to prevent fatal and non-fatal opioid overdoses among female adults released from prison.

DETAILED DESCRIPTION:
ROAR examines implementation of a novel overdose prevention strategy for justice-involved women as they re-enter community treatment settings after incarceration. The ODOC pilot project offers initiation of opioid antagonist treatment prior to release (extended-release naltrexone [XR-NTX]), ongoing support from a Certified Recovery Mentor (CRM), and facilitated entry into community treatment for substance use disorders. Community treatment may include continuation of XR-NTX,or transition to agonist therapy including buprenorphine or methadone, or no medication for opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman (including transgender and non-binary adults assigned to women's housing at CCCF)
* 18 years of age or older with a known release date during the 18-month recruitment period
* Be released to Marion, Multnomah, Clackamas or Washington County, Oregon
* Be willing and able to provide informed consent and HIPAA authorization for medical record abstraction and linkage to state administrative data
* Meet DSM-V (Diagnostic and Statistical Manual) criteria for moderate or severe opioid use disorder
* Be willing to establish ongoing care at the community SUD (substance use disorder) treatment site in county of release
* Be willing to initiate XR-NTX prior to release from incarceration
* Not be currently pregnant and must be willing to take at least one evidence-based measure to avoid becoming pregnant during treatment with XR-NTX

Exclusion Criteria: A participant will be excluded if she

* Has a severe medical, psychiatric, or substance use disorder that, in the opinion of the CCCF Qualified Mental Health Professional (QMHP)or study physician, would make study participation hazardous to the participant, compromise study findings, or prevent the participant from completing the study due to imminent risk of death
* Has another medical condition leading XR-NTX to be contraindicated
* Has chronic pain requiring ongoing pain management with opioid analgesics
* Received methadone or buprenorphine maintenance therapy in the 4 weeks prior to consent
* Has a planned surgery or other procedure within the next 4 weeks that will require opioid analgesia

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study sample is composed of women including transgender and non-binary adults assigned to women's housing at Coffee Creek Correctional Facility.
Study Population: The study will directly recruit incarcerated adult females who meet the DSM-V criteria for moderate or severe opioid use disorder. All participants will have a scheduled release date to Marion, Multnomah, Washington, or Clackamas County, Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Any Opioid Overdose | 6 months after release from incarceration
  This is a binary outcome indicating a fatal or non-fatal opioid-related overdose event

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Waddell, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Department of Corrections, Wilsonville, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waddell EN, Baker R, Hartung DM, Hildebran CJ, Nguyen T, Collins DM, Larsen JE, Stack E; ROAR Protocol Development Team. Reducing overdose after release from incarceration (ROAR): study protocol for an intervention to reduce risk of fatal and non-fatal opioid overdose among women after release from prison. Health Justice. 2020 Jul 10;8(1):18. doi: 10.1186/s40352-020-00113-7. PMID 32651887